CLINICAL TRIAL: NCT02946944
Title: Pilot Randomized Study of the Sidlenafil Efficacy in Combination With Oral Anticoagulants in the Treatment of Patients With Intermediate-high Risk of Pulmonary Embolism
Brief Title: Sidlenafil in Combination With Oral Anticoagulants in Patients With Intermediate-high Risk of Pulmonary Embolism
Acronym: PSCAT
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Meshalkin Research Institute of Pathology of Circulation (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NRICP-45734
Record Dates: First submitted 2016-10-20; First posted 2016-10-27 (Estimated); Last update posted 2016-11-01 (Estimated); Status verified 2016-10

CONDITIONS: Pulmonary Embolism; Intermediate-high Risk; Combination of Oral Anticoagulation Therapy and Sildenafil
Keywords: Pulmonary Embolism; sildenafil; oral anticoagulation therapy
MeSH Terms: conditions — Pulmonary Embolism | interventions — Sildenafil Citrate; apixaban

ARMS (2):
- double drug therapy (Experimental)
  Interventions: Drug: Sildenafil/apixaban
- mono drug therapy (Active Comparator)
  Interventions: Drug: apixaban

INTERVENTIONS:
Drug: Sildenafil/apixaban — After arrival to the emergency department, a series of surveys to determine the risk of death from pulmonary embolism are carried out. Then angiography, tensiometry of SBCC, catheter thrombus fragmentation are scheduled. Then puncture of the right jugular vein is performed. PigTail catheter is inserted via guidewire into the pulmonary artery . Angiography of the pulmonary arteries is performed. Miller index is calculated. Catheter thrombus fragmentation is performed by a PigTail catheter. RV, RA pressures are measured. In the ICU heparin is prescribed (of 1000 units per hour) under the control of PTT (50-75s). The next day patients are randomizaed to assign them into 2 groups. Dual drug therapy is going to be administered to this group (experimental): sildenafil 30mg 3p \ g + 10 mg apixaban 2p \ d for 14 days. On the 7th day MSCT angiography of the pulmonary aretry with contrast and echocardiogram are performed. On the 14th day the controlechocardiogram is performed .
  Arms: double drug therapy
Drug: apixaban — After arrival to the emergency department, a series of surveys to determine the risk of death from pulmonary embolism are carried out. Then angiography, tensiometry of SBCC, catheter thrombus fragmentation are scheduled. Then puncture of the right jugular vein is performed. PigTail catheter is inserted via guidewire into the pulmonary artery . Angiography of the pulmonary arteries is performed. Miller index is calculated. Catheter thrombus fragmentation is performed by a PigTail catheter. RV, RA pressures are measured. In the ICU heparin is prescribed (of 1000 units per hour) under the control of PTT (50-75s). The next day patients are randomizaed to assign them into 2 groups.Mono drug therapy is going to be administered to this group (active comparator): apixaban 10 mg 2p \ d for 14 days. On the 7th day MSCT angiography of the pulmonary aretry with contrast and echocardiogram are performed. On the 14th day the controlechocardiogram is performed .
  Arms: mono drug therapy

SUMMARY:
Pilot randomized study of the sidlenafil efficacy in combination with oral anticoagulants in the treatment of patients with intermediate-high risk of pulmonary embolism

ELIGIBILITY:
Inclusion Criteria:

* pulmonary embolism confirmed by CT scan with contrast, with localization of thrombusa in at least one main or proximal lobar pulmonary artery.
* Right-left ventricular ratio (RV / LV) ≥1 derived from the apical four-chamber view
* Who gave written informed consent to participate in research

Exclusion Criteria:

* Age <18 or >80 years
* Symptoms of pulmonary embolism> 14 days
* Inadequate echocardiographic image quality in the apical four-chamber projection, which limits the measurement of RV / LV ratio
* A significant risk of bleeding
* The administration of thrombolytic drugs within the previous 4 days
* Active bleeding
* Known coagulopathy
* Thrombocytopenia <100,10^9 / l
* Previous use of vitamin K antagonists with an INR> 2.5 at admission
* History of any intracranial or spinal surgery or trauma or intracranial / spinal bleeding
* Intracranial neoplasm
* Arteriovenous malformations or aneurysms
* GIH <3 months
* Cataract Surgery
* Obstetrical manipulation
* Cardiopulmonary resuscitation needed.
* Other invasive procedures <10 days
* Allergy, hypersensitivity, thrombocytopenia to heparin or tissue plasminogen activator
* Allergy to iodine contrast
* A well-known right-left cardiac shunt, for example, a large patent foramen ovale, or atrial septal defect; large (> 10 mm), or a blood clot in right atrium/right ventricle
* Systolic blood pressure <90 mm Hg for at least 15 minutes, or fall of systolic blood pressure is not less than 40 mm Hg for at least 15 min., with evidence of organ hypoperfusion (cold extremities or low diuresis <30 mL / h, or confusion), or the need for administration of catecholamines to maintain adequate perfusion of organs and systolic blood pressure> 90 mm Hg
* Severe hypertension (systolic> 180 mm Hg or diastolic> 105 mm Hg.).
* Pregnancy, lactation, delivery<30 days
* Participation in any other study (drug or device)
* Life expectancy <90 days
* Refusal to participate in the study

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2016-10; Primary Completion 2020-10 (Estimated); Study Completion 2020-10 (Estimated)

PRIMARY OUTCOMES:
MSCT RV \ LV Index | 7th day
  on the 7th day of treatment RV \ LV Index (calculated according to MSCT angiography of the pulmonary arteries)

SECONDARY OUTCOMES:
Echocardiogram RV \ LV Index | 7th day
  Echocardiogram (an index of RV \ LV) on 7th day
Echocardiogram RV \ LV Index | 14th day
  Echocardiogram (an index of RV \ LV) on 14th day
Echocardiogram RV \ LV Index | one month
  Echocardiogram (an index of RV \ LV) on one month
Echocardiogram pressure in the pulmonary artery | one month
  the average pressure in the pulmonary artery according to echocardiography
hemodynamic instability | one month
  in the hospital and within a month follow-up
death | one month
  in the hospital and within a month follow-up
bleeding | one month
  clinically significant bleeding on a scale HAS-BLED
recurrent venous thrombosis | one month
  recurrent venous thrombosis
recurrent pulmonary embolism | one month
  recurrent pulmonary embolism.

CONTACTS AND LOCATIONS:
Locations (1):
- Federal State Institution Academician E.N.Meshalkin Novosibirsk State Research Institute Of Circulation Pathology Rusmedtechnology, Novosibirsk, Russia